CLINICAL TRIAL: NCT00202644
Title: A Phase IIIb, Randomized, Open Label Study to Compare the Safety, Efficacy and Tolerability of Anagrelide Hydrochloride Versus Hydroxyurea in High-Risk Essential Thrombocythaemia Patients.
Brief Title: A Study of Anagrelide and Hydroxyurea in High-Risk Essential Thrombocythemia Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPD422-403; 2004-004061-15 (EudraCT Number)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2018-01-24 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Thrombocythemia, Hemorrhagic
MeSH Terms: conditions — Thrombocythemia, Essential | interventions — anagrelide; Hydroxyurea

ARMS (2):
- A (Experimental)
  Interventions: Drug: Anagrelide
- B (Active Comparator)
  Interventions: Drug: Hydroxyurea

INTERVENTIONS:
Drug: Anagrelide — Anagrelide hydrochloride 0.5mg capsules;initial dose administered will be 1.0mg/day administered as 0.5mg bid. The dose will be titrated such that the total daily dose is incremented by no more than 0.5mg per week as required depending on platelet reduction versus adverse event profile.
  Arms: A
Drug: Hydroxyurea — Hydroxyurea is 500mg hydroxycarbamide capsules; initial dose is 1000mg/day, administered in two divided doses (500mg/dose). Dose titrated to effect to achieve a response.
  Arms: B

SUMMARY:
Essential thrombocythaemia is a disorder of bone marrow, which causes too many platelets to be produced. Platelets are small cells carried around in the blood, which help form blood clots. When patients have too many platelets, there is a risk of blood clots forming unnecessarily and excessive bleeding. The aim of this study is to gain additional information on the safety profile of Anagrelide (Xagrid(r)) and Hydroxyurea (also known as hydroxycarbamide).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of essential thrombocythaemia - high risk profile
* Previously untreated with a cytoreductive agent
* Females of childbearing potential must have a negative urine pregnancy test prior to entering the study and must agree to use effective birth control for the duration of the study

Exclusion Criteria:

* Diagnosis of any other myeloproliferative disorder
* Any known cause for a secondary thrombocytosis
* Anti-coagulant and anti-aggregant therapies
* Known or suspected heart disease
* Left Ventricular Ejection Fraction < 55%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2006-01-13 (Actual); Primary Completion 2015-12-15 (Actual); Study Completion 2015-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (15):
- Bulgaria (3):
  - University Multiprofile Hospital for Active Treatment ''Dr Georgi Stranski'' - Pleven, Pleven
  - University Multiprofile Hospital for active Treatment ''Alexandrovska'' Clinic of Haematology, Sofia
  - University Multiprofile Hospital for Active Treament ''Sv. Marina'' - Varna Haematology Clinic, Varna
- France (2):
  - CHU Angers Services des Maladies du Sang, Angers, Cedex 09
  - Hopital Saint Louis - Centre d'Investigation Clinique, Paris
- Hungary (4):
  - University of Debrecen Medical and Health Science Centre, Debrecen
  - Petz Aladar County Teaching Hospital, Győr
  - Pandy Kalman Hospital of Bekes County, Gyula
  - Kaposi Mor Teaching Hospital, Kaposvár
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne Katedra i Klinika Hematologii i Transplantologii, Gdansk
  - Samodzielny Publiczny Szpital Kliniczny Nr 1, Lublin
  - Katedra i Klinika Onkologii i Chorob Wewnetrznych Akademii Medycznej, Warsaw
  - Klinika Hematologii Instytut Hematologii i Transfuzjologi, Warsaw
- Hospitals da Universidade de Coimbra, Coimbra, Portugal
- Institute for Haematology of Clinical Centre of Serbia, Belgrade, Serbia

REFERENCES:
- [Result] Birgegard G, Folkvaljon F, Garmo H, Holmberg L, Besses C, Griesshammer M, Gugliotta L, Wu J, Achenbach H, Kiladjian JJ, Harrison CN. Leukemic transformation and second cancers in 3649 patients with high-risk essential thrombocythemia in the EXELS study. Leuk Res. 2018 Nov;74:105-109. doi: 10.1016/j.leukres.2018.10.006. Epub 2018 Oct 11. PMID 30368038
- [Derived] Gotic M, Egyed M, Gercheva L, Warzocha K, Kvasnicka HM, Achenbach H, Wu J. Cardiovascular Safety of Anagrelide Hydrochloride versus Hydroxyurea in Essential Thrombocythaemia. Cardiovasc Toxicol. 2021 Mar;21(3):236-247. doi: 10.1007/s12012-020-09615-0. Epub 2020 Oct 29. PMID 33123978

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 183 participants were screened, 149 participants were randomized at 29 sites across 10 countries. Four (4) participants randomized but withdrawn prior to treatment and 1 participant not randomized but treated.
Groups:
- Anagrelide: Participants received Anagrelide hydrochloride 1.0 milligram (mg) per day administered orally as 0.5 mg capsule twice daily (bid) for 1 week. Then the dose was titrated such that the total daily dose is incremented by no more than 0.5 mg in any 1 week and the recommended maximum single dose could not exceed 2.5 mg as required depending on platelet reduction versus adverse event profile. Total daily dosage was not exceed 10 mg. Participants followed for up to 3 years.
- Hydroxyurea: Participants received Hydroxyurea as 1000 mg per day administered orally as 500 mg capsule twice daily and dose titrated to effect to achieve a response. Participants followed for up to 3 years.
Period: Overall Study
Arm/Group | Anagrelide | Hydroxyurea
Started | 76 (One participant not randomized but treated.) | 70
Completed | 41 | 43
Not Completed | 35 | 27
Not completed — Adverse Event | 12 | 13
Not completed — Withdrawal by Subject | 8 | 6
Not completed — Lack of Efficacy | 6 | 6
Not completed — Lost to Follow-up | 0 | 1
Not completed — Other | 9 | 1

BASELINE CHARACTERISTICS:
Population: The safety population was defined as all participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Anagrelide | Hydroxyurea | Total
Number analyzed (Participants) | 76 | 70 | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (16.10) | 52.9 (15.80) | 52.5 (15.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 45 | 101
  Male | 20 | 25 | 45

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Left Ventricular Ejection Fraction (LVEF) Over Time
Description: The LVEF was measured by echocardiography and considered a sufficiently sensitive measure to evaluate any changes in cardiac function.
Time Frame: Baseline and Month 1, 2, 3, 6, 9, 12, 18, 24, 30 and 36
Population: The Full Analysis Set (FAS) population included all randomized participants who received at least 1 dose of study medication and who had a pretreatment and at least 1 post baseline LVEF measurement recorded. Here, n = Number of participants analysed for specified category at the specified time points in each arm respectively.
Measure: Mean (Standard Deviation); unit: percentage of ejection fraction
Arm/Group | Anagrelide | Hydroxyurea
Number analyzed (Participants) | 73 | 68
percentage of ejection fraction
  Baseline | 66.4 (4.81) | 66.9 (4.59)
  Change from baseline at Month 1: number analyzed (Participants) | 71 | 64
  Change from baseline at Month 1 | 0.5 (4.68) | -1.1 (4.73)
  Change from baseline at Month 2: number analyzed (Participants) | 68 | 63
  Change from baseline at Month 2 | 1.2 (5.80) | 0 (5.03)
  Change from baseline at Month 3: number analyzed (Participants) | 67 | 62
  Change from baseline at Month 3 | 0.1 (5.31) | -0.4 (3.94)
  Change from baseline at Month 6: number analyzed (Participants) | 59 | 60
  Change from baseline at Month 6 | -0.5 (5.68) | -0.6 (3.95)
  Change from baseline at Month 9: number analyzed (Participants) | 52 | 52
  Change from baseline at Month 9 | -0.8 (4.78) | -1.5 (5.15)
  Change from baseline at Month 12: number analyzed (Participants) | 45 | 52
  Change from baseline at Month 12 | -0.8 (6.61) | -0.6 (5.67)
  Change from baseline at Month 18: number analyzed (Participants) | 41 | 48
  Change from baseline at Month 18 | -2.0 (5.54) | -1.2 (4.84)
  Change from baseline at Month 24: number analyzed (Participants) | 40 | 49
  Change from baseline at Month 24 | -1.8 (6.81) | -1.7 (6.17)
  Change from baseline at Month 30: number analyzed (Participants) | 40 | 45
  Change from baseline at Month 30 | -1.8 (5.84) | -0.2 (5.38)
  Change from baseline at Month 36: number analyzed (Participants) | 40 | 44
  Change from baseline at Month 36 | -1.7 (6.55) | -0.6 (5.46)

2. Primary Outcome: Platelet Count at Month 6
Description: Platelet count was evaluated.
Time Frame: Month 6
Population: The FAS population included all randomized participants who received at least 1 dose of study medication and who had a pretreatment and at least 1 post baseline LVEF measurement recorded. Here, N = Number of participants analysed in each arm for this outcome measure.
Measure: Mean (Standard Deviation); unit: 10^9 platelets per liter
Arm/Group | Anagrelide | Hydroxyurea
Number analyzed (Participants) | 60 | 58
10^9 platelets per liter | 418.6 (135.96) | 396.0 (144.07)
Statistical Analysis 1: Comparison: Anagrelide vs Hydroxyurea; Test type: Non-Inferiority or Equivalence — Noninferiority of anagrelide could be concluded if lower limit of 95% Confidence Interval for the difference between treatment groups (Hydroxyurea - Anagrelide) was > -100 x 10^9/Liter; Least Square Mean = -100.5, 95% CI 2-sided [-179.42 to -21.49], Standard Error of Mean 39.93

3. Secondary Outcome: Change From Baseline in Platelet Counts at Month 3 and 36
Description: Platelet count was evaluated throughout the study.
Time Frame: Baseline and Month 3 and 36
Population: The FAS population included all randomized participants who received at least 1 dose of study medication and who had a pretreatment and at least 1 post baseline LVEF measurement recorded with last observation carried forward (LOCF). Here, n=number of participants analysed for specified category at specified time points in each arm respectively.
Measure: Mean (Standard Deviation); unit: 10^9 platelets per liter
Arm/Group | Anagrelide | Hydroxyurea
Number analyzed (Participants) | 73 | 68
10^9 platelets per liter
  Change from baseline at Month 3 | 575.3 (36.11) | 462.2 (37.54)
  Change from baseline at Month 36 | 531.0 (42.14) | 462.8 (43.81)
Statistical Analysis 1: Comparison: Anagrelide vs Hydroxyurea; Month 3; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Least Square Mean = -113.1, 95% CI 2-sided [-187.40 to -38.83], Standard Error of Mean 37.56
Statistical Analysis 2: Comparison: Anagrelide vs Hydroxyurea; Month 36; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Least Square Mean = -68.3, 95% CI 2-sided [-154.95 to 18.43], Standard Error of Mean 43.83

4. Secondary Outcome: Percentage of Participants With Complete Response
Description: A complete response was defined as a platelet count of less than (<) 400x10^9/Liter which was confirmed over 2 consecutive visits at least 28 days apart.
Time Frame: Baseline up to Month 36
Population: The FAS population included all randomized participants who received at least 1 dose of study medication and who had a pretreatment and at least 1 post baseline LVEF measurement recorded.
Measure: Number; unit: percenatge of participants
Arm/Group | Anagrelide | Hydroxyurea
Number analyzed (Participants) | 73 | 68
percenatge of participants | 58.9 | 58.8

5. Secondary Outcome: Percentage of Participants With Partial Response
Description: A partial response is defined as a platelet count of 400-600 x 10^9/Liter and a reduction in platelet count of at least 200 x 10^9/Liter from baseline which was confirmed over 2 consecutive visits at least 28 days apart.
Time Frame: Baseline up to Month 36
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Anagrelide | Hydroxyurea
Number analyzed (Participants) | 73 | 68
percentage of participants | 21.9 | 27.9

6. Secondary Outcome: Time to Complete Response
Description: Time in days from the date of the first dose of study medication to the date of the first visit at which response was classified. If a participant did not achieve response then they were censored at their last visit in the study (Month 36 or withdrawal).
Time Frame: Baseline up to Month 36
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Anagrelide | Hydroxyurea
Number analyzed (Participants) | 73 | 68
days | 177.0 [129.0 to 548.0] | 123.0 [90.0 to 554.0]

7. Secondary Outcome: Time to Partial Response
Description: as for outcome 6
Time Frame: Baseline up to Month 36
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Anagrelide | Hydroxyurea
Number analyzed (Participants) | 73 | 68
days | 61.0 [43.0 to 85.0] | 47.0 [41.0 to 57.0]

8. Secondary Outcome: Number of Participants With Thrombotic and Haemorrhagic Events
Description: Thrombohaemorrhagic events are a well-known complication of the underlying essential thrombocythemia (ET) and disease progression. Events such as arterial and venous thrombosis, serious haemorrhage (including gastrointestinal haemorrhage), and death from vascular causes have been reported in participants who received cytoreductive treatment.
Time Frame: From the signing of informed consent until the last study-related visit (Month 36)
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Anagrelide | Hydroxyurea
Number analyzed (Participants) | 73 | 68
participants | 30 | 16

9. Secondary Outcome: Change From Baseline in White Blood Cell Count Over Time
Description: White blood cell count was evaluated throughout the study.
Time Frame: Baseline and Month 6, 12, 18, 24, 30 and 36
Population: The FAS population included all randomized participants who received at least 1 dose of study medication and who had a pretreatment and at least 1 post baseline LVEF measurement recorded. Here, n = Number of participants analysed for specified category at the specified time points in each arm respectively.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Anagrelide | Hydroxyurea
Number analyzed (Participants) | 73 | 68
10^9 cells per liter
  Baseline | 9.13 (2.159) | 10.20 (3.491)
  Change from baseline at Month 6: number analyzed (Participants) | 60 | 58
  Change from baseline at Month 6 | -0.38 (4.257) | -5.02 (2.525)
  Change from baseline at Month 12: number analyzed (Participants) | 45 | 51
  Change from baseline at Month 12 | -1.00 (2.001) | -4.79 (2.779)
  Change from baseline at Month 18: number analyzed (Participants) | 42 | 49
  Change from baseline at Month 18 | -1.18 (2.184) | -4.46 (2.664)
  Change from baseline at Month 24: number analyzed (Participants) | 40 | 49
  Change from baseline at Month 24 | -1.24 (2.283) | -4.82 (2.692)
  Change from baseline at Month 30: number analyzed (Participants) | 40 | 45
  Change from baseline at Month 30 | -1.00 (2.316) | -4.59 (3.391)
  Change from baseline at Month 36: number analyzed (Participants) | 40 | 43
  Change from baseline at Month 36 | -1.63 (2.234) | -4.46 (3.312)

10. Secondary Outcome: Change From Baseline in Red Blood Cell Count Over Time
Description: Red blood cell count was evaluated throughout the study.
Time Frame: Baseline and Month 6, 12, 18, 24, 30 and 36
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Anagrelide | Hydroxyurea
Number analyzed (Participants) | 73 | 68
10^12 cells per liter
  Baseline | 4.757 (0.5897) | 4.787 (0.6002)
  Change from baseline at Month 6: number analyzed (Participants) | 60 | 58
  Change from baseline at Month 6 | -0.227 (0.4134) | -1.467 (0.6563)
  Change from baseline at Month 12: number analyzed (Participants) | 45 | 51
  Change from baseline at Month 12 | -0.246 (0.4292) | -1.398 (0.5744)
  Change from baseline at Month 18: number analyzed (Participants) | 42 | 49
  Change from baseline at Month 18 | -0.225 (0.4224) | -1.323 (0.7278)
  Change from baseline at Month 24: number analyzed (Participants) | 40 | 49
  Change from baseline at Month 24 | -0.299 (0.5811) | -1.281 (0.7219)
  Change from baseline at Month 30: number analyzed (Participants) | 40 | 45
  Change from baseline at Month 30 | -0.295 (0.5713) | -1.339 (0.6509)
  Change from baseline at Month 36: number analyzed (Participants) | 40 | 43
  Change from baseline at Month 36 | -0.366 (0.4328) | -1.362 (0.6586)

ADVERSE EVENTS:
Time Frame: From the signing of informed consent until the last study-related visit (Month 36)
Arm/Group | Anagrelide | Hydroxyurea
Serious Adverse Events (participants affected / at risk) | 17/76 | 13/70
Other Adverse Events (participants affected / at risk) | 46/76 | 27/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anagrelide (N=76) | Hydroxyurea (N=70)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (2)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic amputation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendon calcification (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adenoid cystic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Peripheral nerve sheath tumour malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (2) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 3 (3) | 0 (0)
Neurological decompensation (Nervous system disorders) | 1 (1) | 0 (0)
Vasculitis cerebral (Nervous system disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anagrelide (N=76) | Hydroxyurea (N=70)
Anaemia (Blood and lymphatic system disorders) | 4 (6) | 8 (9)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 7 (7)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 5 (8)
Palpitations (Cardiac disorders) | 18 (29) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 5 (5) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (7) | 3 (3)
Asthenia (General disorders) | 5 (6) | 4 (6)
Chest pain (General disorders) | 4 (7) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 5 (8)
Pharyngitis (Infections and infestations) | 2 (2) | 6 (8)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (8) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 2 (2)
Headache (Nervous system disorders) | 19 (33) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2)
Hypertension (Vascular disorders) | 9 (12) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.